CLINICAL TRIAL: NCT04541186
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Explore the Efficacy and Safety of BIO89-100 in Subjects With Severe Hypertriglyceridemia
Brief Title: Study to Explore the Efficacy and Safety of BIO89-100 (Pegozafermin) in Participants With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO89-100-221
Record Dates: First submitted 2020-08-14; First posted 2020-09-09 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: Severe Hypertriglyceridemia
Keywords: Hypertriglyceridemia; Dyslipidemia; Lipid disorder; FGF21
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Pegozafermin 9 mg QW (Experimental): Participants received pegozafermin 9 mg QW as an SC injection for 8 weeks in the Main Study cohort.
  Interventions: Drug: Pegozafermin
- Pegozafermin 18 mg QW (Experimental): Participants received pegozafermin 18 mg QW as an SC injection for 8 weeks in the Main Study cohort.
  Interventions: Drug: Pegozafermin
- Pegozafermin 27 mg QW (Experimental): Participants received pegozafermin 27 mg QW as an SC injection for 8 weeks in the Main Study cohort or Fibrate Expansion cohort. Main Study and Fibrate Expansion pegozafermin 27 mg QW groups were pooled together due to low sample size in the expansion cohort.
  Interventions: Drug: Pegozafermin
- Pegozafermin 36 mg Q2W (Experimental): Participants received pegozafermin 36 mg Q2W as an SC injection for 8 weeks in the Main Study cohort.
  Interventions: Drug: Pegozafermin
- Placebo (Placebo Comparator): Matching placebo was injected at matching frequency per assigned cohort for 8 weeks in the Main Study cohort or Fibrate Expansion cohort. Main Study and Fibrate Expansion placebo groups were pooled together due to low sample size in the expansion cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pegozafermin — Subcutaneous injection
  Other Names: BIO89-100
  Arms: Pegozafermin 18 mg QW; Pegozafermin 27 mg QW; Pegozafermin 36 mg Q2W; Pegozafermin 9 mg QW
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy, safety, and tolerability of different doses and dose regimens (once weekly [QW] or every 2 weeks [Q2W]), subcutaneous (SC) dosing of BIO89-100 (pegozafermin) compared to placebo in participants with severe hypertriglyceridemia (SHTG).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥21 to ≤75 years.
2. Screening fasting triglyceride ≥500 milligrams (mg)/deciliters (dL) and ≤2000 mg/dL.
3. Willing to maintain current eating and exercise habits from time of signing the informed consent and for the duration of the study.
4. Participants could be taking statins and/or prescription fish oil as background therapy or not be taking any background therapy.
5. Magnetic resonance imaging - whole liver proton density fat fraction (MRI-PDFF) of ≥6% for participants screened for the Fibrate Expansion cohort.

Exclusion Criteria:

1. Uncontrolled or newly diagnosed hypertension.
2. Body mass index >45 kilograms (kg)/meters squared (m^2).
3. Receiving niacin, proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors, or supplements that could lower lipid levels.
4. Type 1 diabetes mellitus.
5. Diagnosis of Type 2 diabetes mellitus <6 months prior to screening.
6. History of malignancy within 5 years prior to screening.
7. Participants with known lipoprotein lipase impairment or deficiency (Fredrickson Type 1), apolipoprotein C-II deficiency, or familial dysbetalipoproteinemia (Fredrickson Type 3).
8. Clinically or otherwise documented cardiovascular or cerebrovascular disease.
9. Weight change ≥5% in 3 months prior to first screening visit or weight change ≥5% during screening or planning to try to lose weight during conduct of study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (29):
  - 89Bio Clinical Study Site, La Mesa, California
  - 89Bio Clinical Study Site, San Francisco, California
  - 89Bio Clinical Study Site, Clearwater, Florida
  - 89Bio Clinical Study Site, Greenacres City, Florida
  - 89Bio Clinical Study Site, Jacksonville, Florida
  - 89Bio Clinical Study Site, Miami, Florida
  - 89Bio Clinical Study Site, Miami Lakes, Florida
  - 89Bio Clinical Study Site, North Miami Beach, Florida
  - 89Bio Clinical Study Site, Orlando, Florida
  - 89Bio Clinical Study Site, Tampa, Florida
  - 89Bio Clinical Study Site, Lawrenceville, Georgia
  - 89Bio Clinical Study Site, Quincy, Illinois
  - 89Bio Clinical Study Site, Wauconda, Illinois
  - 89Bio Clinical Study Site, West Des Moines, Iowa
  - 89Bio Clinical Study Site, Louisville, Kentucky
  - 89Bio Clinical Study Site, Olive Branch, Mississippi
  - 89Bio Clinical Study Site, Albany, New York
  - 89Bio Clinical Study Site, Greensboro, North Carolina
  - 89Bio Clinical Study Site, Morganton, North Carolina
  - 89Bio Clinical Study Site, Marion, Ohio
  - 89Bio Clinical Study Site, Summerville, South Carolina
  - 89Bio Clinical Study Site, Chattanooga, Tennessee
  - 89Bio Clinical Study Site, Kingsport, Tennessee
  - 89Bio Clinical Study Site, Austin, Texas
  - 89Bio Clinical Study Site, Dallas, Texas
  - 89Bio Clinical Study Site, Houston, Texas
  - 89Bio Clinical Study Site, Lampasas, Texas
  - 89Bio Clinical Study Site, Magnolia, Texas
  - 89Bio Clinical Study Site, Manassas, Virginia
- Czechia (2):
  - 89Bio Clinical Study Site, Pardubice
  - 89Bio Clinical Study Site, Prague
- Hungary (5):
  - 89Bio Clinical Study Site, Miskolc, Borsod-Abauj Zemplen county
  - 89Bio Clinical Study Site, Baja
  - 89Bio Clinical Study Site, Békéscsaba
  - 89Bio Clinical Study Site, Budapest
  - 89Bio Clinical Study Site, Debrecen
- Poland (5):
  - 89Bio Clinical Study Site, Bialystok
  - 89Bio Clinical Study Site, Lodz
  - 89Bio Clinical Study Site, Oświęcim
  - 89Bio Clinical Study Site, Rzeszów
  - 89Bio Clinical Study Site, Torun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhatt DL, Bays HE, Miller M, Cain JE 3rd, Wasilewska K, Andrawis NS, Parli T, Feng S, Sterling L, Tseng L, Hartsfield CL, Agollah GD, Mansbach H, Kastelein JJP; ENTRIGUE Principal Investigators. The FGF21 analog pegozafermin in severe hypertriglyceridemia: a randomized phase 2 trial. Nat Med. 2023 Jul;29(7):1782-1792. doi: 10.1038/s41591-023-02427-z. Epub 2023 Jun 24. PMID 37355760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per the Statistical Analysis Plan (SAP), since a low number of participants enrolled in the fibrate cohort (3 on placebo and 3 on active treatment [pegozafermin]), participants in the pegozafermin 27 mg QW fibrate cohort were combined with the pegozafermin 27 mg QW main cohort, forming a pooled pegozafermin 27 mg QW group for analyses. Similarly, the placebo participants in the fibrate cohort were combined with the main placebo group (pooled) for analyses.
Groups:
- Pegozafermin 9 mg QW: Pegozafermin 9 mg QW was administered as a subcutaneous (SC) injection.
- Pegozafermin 18 mg QW: Pegozafermin 18 mg QW was administered as an SC injection.
- Pegozafermin 27 mg QW: Pegozafermin 27 mg QW was administered as an SC injection.
- Pegozafermin 36 mg Q2W: Pegozafermin 36 mg Q2W was administered as an SC injection.
- Placebo: Matching placebo was injected at matching frequency per assigned cohort.
Period: Main Study
Arm/Group | Pegozafermin 9 mg QW | Pegozafermin 18 mg QW | Pegozafermin 27 mg QW | Pegozafermin 36 mg Q2W | Placebo
Started (Randomization set summarized based on planned treatment.) | 16 | 17 | 16 | 16 | 15
Safety Analysis Set (Participants who received at least 1 dose of study drug. Safety Analysis Set is summarized based treatment received.) | 12 (4 participants randomized to receive 9 mg QW received 18 mg QW instead) | 21 (4 participants randomized to receive 9 mg QW received 18 mg QW instead) | 15 | 16 | 15
Full Analysis Set (FAS) (Participants who received at least 1 dose of study drug, had a baseline, and at least 1 post-baseline triglyceride measurement not including end of study (EOS) visit.) | 16 | 17 | 13 | 16 | 14
Completed | 15 | 16 | 10 | 15 | 14
Not Completed | 1 | 1 | 6 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 4 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — COVID-19-related Dose Interruption | 0 | 0 | 0 | 0 | 1
Not completed — Randomized in Error Not Treated | 0 | 0 | 1 | 0 | 0
Period: Fibrate Expansion Study
Arm/Group | Pegozafermin 9 mg QW | Pegozafermin 18 mg QW | Pegozafermin 27 mg QW | Pegozafermin 36 mg Q2W | Placebo
Started | 0 | 0 | 3 | 0 | 3
Received at Least 1 Dose of Study Drug | 0 | 0 | 3 | 0 | 3
Full Analysis Set (Participants who received at least 1 dose of study drug, had a baseline, and at least 1 post-baseline TG measurement not including EOS visit.) | 0 | 0 | 3 | 0 | 3
Completed | 0 | 0 | 3 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Other than Specified | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug. Participants are summarized by treatment received.
  As per SAP, since a low number of participants enrolled in the fibrate cohort, participants randomized to pegozafermin 27 mg QW fibrate cohort were combined with the pegozafermin 27 mg QW main cohort, forming a pooled pegozafermin 27 mg QW group for analyses. Similarly, the placebo participants in the fibrate cohort were combined with the main placebo group.
Groups:
- Pegozafermin 9 mg QW: Pegozafermin 9 mg QW was administered as a SC injection.
- Pegozafermin 27 mg QW: Pegozafermin 27 mg QW was administered as an SC injection. The Main Study cohort and Fibrate Expansion cohort for pegozafermin 27 mg were pooled together due to low sample size in the expansion cohort.
- Placebo: Matching placebo was injected at matching frequency per assigned cohort. Main Study cohort and Fibrate Expansion cohort for placebo were pooled together due to low sample size in the expansion cohort.
- Total: Total of all reporting groups
Arm/Group | Pegozafermin 9 mg QW | Pegozafermin 18 mg QW | Pegozafermin 27 mg QW | Pegozafermin 36 mg Q2W | Placebo | Total
Number analyzed (Participants) | 12 | 21 | 18 | 16 | 18 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.12) | 51.3 (10.81) | 53.9 (7.18) | 53.1 (12.36) | 57.5 (10.30) | 53.7 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 2 | 6 | 21
  Male | 8 | 17 | 13 | 14 | 12 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 5 | 3 | 17
  Not Hispanic or Latino | 9 | 19 | 14 | 11 | 15 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 1 | 0 | 0 | 0 | 1 | 2
  Race: White | 11 | 21 | 18 | 14 | 17 | 81
  Race: Not Reported | 0 | 0 | 0 | 1 | 0 | 1
  Race: Unknown | 0 | 0 | 0 | 1 | 0 | 1
Triglyceride (TG) Level [Count of Participants; unit: Participants]
  <750 mg/dL | 9 | 14 | 12 | 9 | 13 | 57
  ≥750 mg/dL | 3 | 7 | 6 | 7 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 8 in Serum Triglyceride (TG)
Time Frame: Baseline, Week 8
Population: FAS: Participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline TG measurement not including EOS visit. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. As pre-specified in the SAP, the sample size in each arm (by dose group) was insufficient (under powered) to effectively evaluate differences in efficacy by dose, therefore, efficacy analysis was performed using total pegozafermin and placebo groups.
Measure: Median (Inter-Quartile Range); unit: percent change from Baseline
Groups:
- Pegozafermin: All participants who were randomized to pegozafermin in the main study and fibrate expansion cohort were pooled together.
- Placebo: Participants randomized to placebo in the main study and fibrate expansion cohort were pooled together.
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 64 | 17
percent change from Baseline | -57.33 [-69.07 to -32.31] | -11.85 [-23.22 to 7.88]
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; Test type: Superiority; p < 0.001, van Elteren test — Significant level = 0.05; Nonparametric analysis stratified by baseline TG level and background lipid therapy to test the treatment difference using pooled data; Median Percent Change Difference = -43.73, 95% CI 2-sided [-57.08 to -30.31] — The location shift and Hodges-Lehmann 95% confidence interval were based on Hodges-Lehman estimation. Placebo group is the reference group, and the comparison was performed in pooled pegozafermin treatment group vs. placebo pooled

2. Secondary Outcome: Number of Participants Who Achieved TG <500 mg/dL at Week 8
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 64 | 17
Participants | 51 | 5
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Significant level = 0.05; Cochran-Mantel-Haenszel test stratified by baseline TG level and lipid modifying therapy use

3. Secondary Outcome: Percent Change From Baseline to Week 8 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C), Apolipoprotein B100 (ApoB), Low-density Lipoprotein Cholesterol (LDL-C), and High-density Lipoprotein Cholesterol (HDL-C)
Description: Least Squares Means were calculated using mixed-model repeated measures (MMRM).
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 63 | 17
percent change from Baseline
  Non-HDL-C | -18.29 (2.943) | -0.57 (5.586)
  ApoB | -10.51 (2.238) | 1.07 (4.309)
  LDL-C: number analyzed (Participants) | 62 | 15
  LDL-C | 10.44 (4.654) | 8.72 (9.018)
  HDL-C | 24.65 (3.752) | 9.67 (7.045)
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; MMRM analysis of non-HDL-C comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.007, MMRM — Significant level = 0.05; Least Squares Means Difference = -17.87, 95% CI 2-sided [-30.67 to -5.07], Standard Error of Mean 6.425
Statistical Analysis 2: Comparison: Pegozafermin vs Placebo; MMRM analysis of ApoB comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.019, MMRM — Significant level of 0.05; Least Squares Means Difference = -11.75, 95% CI 2-sided [-21.48 to -2.01], Standard Error of Mean 4.888
Statistical Analysis 3: Comparison: Pegozafermin vs Placebo; MMRM analysis of LDL-C comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.870, MMRM — Significant level = 0.05; Least Squares Means Difference = 1.73, 95% CI 2-sided [-19.21 to 22.68], Standard Error of Mean 10.519
Statistical Analysis 4: Comparison: Pegozafermin vs Placebo; MMRM analysis of HDL-C comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.064, MMRM — Significant level = 0.05; Least Squares Means Difference = 15.41, 95% CI 2-sided [-0.89 to 31.70], Standard Error of Mean 8.182

4. Secondary Outcome: Percent Change From Baseline to Week 8 in Very Low-density Lipoprotein Cholesterol (VLDL-C) and VLDL-TG
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 62 | 15
percent change from Baseline
  VLDL-C | -47.96 [-63.14 to -16.67] | -0.41 [-30.38 to 10.98]
  VLDL-TG: number analyzed (Participants) | 61 | 15
  VLDL-TG | -58.50 [-72.53 to -32.80] | -0.85 [-27.72 to 14.25]
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; Nonparametric analysis of VLDL-C comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.006, van Elteren Test — Significant level = 0.05
Statistical Analysis 2: Comparison: Pegozafermin vs Placebo; Nonparametric analysis of VLDL-TG comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.002, van Elteren test — Significant level of 0.05

5. Secondary Outcome: Percent Change in Baseline to Week 8 in Fasting Plasma Glucose, Adiponectin, and Body Weight
Description: Least Squares Mean was calculated using MMRM.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 63 | 17
percent change from Baseline
  Fasting Plasma Glucose | -3.90 (2.681) | -2.67 (5.230)
  Adiponectin | 69.53 (7.383) | 5.70 (14.556)
  Body Weight | -0.15 (0.339) | -0.14 (0.654)
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; MMRM analysis of fasting plasma glucose comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.809, MMRM — Significant level = 0.05
Statistical Analysis 2: Comparison: Pegozafermin vs Placebo; MMRM analysis of adiponectin comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p < 0.001, MMRM — Significant level = 0.05
Statistical Analysis 3: Comparison: Pegozafermin vs Placebo; MMRM analysis of body weight comparison between pegozafermin pooled versus placebo pooled group; Test type: Superiority; p = 0.973, MMRM — Significant level = 0.05

6. Secondary Outcome: Percent Change From Baseline to Week 8 in Liver Fat as Assessed by Magnetic Resonance Imaging - Whole Liver Proton Density Fat Fraction (MRI-PDFF)
Description: Least Squares Mean was calculated using analysis of covariance (ANCOVA).
Time Frame: Baseline, Week 8
Population: All participants in the FAS who had baseline and a follow-up MRI-PDFF assessment. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. As pre-specified in the SAP, the sample size in each arm (by dose group) was insufficient (under powered) to effectively evaluate differences in efficacy by dose, therefore, efficacy analysis was performed using total pegozafermin and placebo groups.
Measure: Least Squares Mean (Standard Error); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 17 | 6
percent change from Baseline | -42.18 (6.207) | -8.26 (11.214)
Statistical Analysis 1: Comparison: Pegozafermin vs Placebo; Test type: Superiority; p = 0.012, ANCOVA — Significant level = 0.05

7. Secondary Outcome: Percent Change From Baseline to Week 8 in High-sensitivity C-reactive Protein (hsCRP)
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 63 | 17
percent change from Baseline | -21.43 [-43.30 to 42.37] | -1.10 [-50.41 to 18.84]

8. Secondary Outcome: Percent Change From Baseline to Week 8 in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Least Squares Mean was calculated using MMRM.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from Baseline
Arm/Group | Pegozafermin | Placebo
Number analyzed (Participants) | 63 | 17
percent change from Baseline
  ALT | -4.28 (4.549) | 0.43 (8.881)
  AST | -11.50 (3.341) | 0.51 (6.597)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to 12 weeks
Description: As per the SAP, since a low number of participants enrolled in the fibrate cohort, participants in the pegozafermin 27 mg QW fibrate cohort were pooled with the pegozafermin 27 mg QW main cohort. Similarly, placebo groups in main and fibrate cohorts were pooled.
  Safety Analysis Set: Participants who received at least 1 dose of study drug. Safety data analysis was by treatment group received. 4 participants randomized to receive 9 mg QW received 18 mg QW instead.
Arm/Group | Pegozafermin 9 mg QW | Pegozafermin 18 mg QW | Pegozafermin 27 mg QW | Pegozafermin 36 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/21 | 0/18 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/21 | 1/18 | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 7/12 | 13/21 | 13/18 | 7/16 | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegozafermin 9 mg QW (N=12) | Pegozafermin 18 mg QW (N=21) | Pegozafermin 27 mg QW (N=18) | Pegozafermin 36 mg Q2W (N=16) | Placebo (N=18)
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegozafermin 9 mg QW (N=12) | Pegozafermin 18 mg QW (N=21) | Pegozafermin 27 mg QW (N=18) | Pegozafermin 36 mg Q2W (N=16) | Placebo (N=18)
Injection site reaction (General disorders) | 1 | 2 | 1 | 2 | 0
Injection site erythema (General disorders) | 0 | 1 | 2 | 1 | 0
Injection site pruritus (General disorders) | 1 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 3 | 0 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 2
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study did not separately evaluate the response to pegozafermin in participants who were on and who were not on concurrent fibrate therapy due to small sample size in the Fibrate Expansion cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT04541186/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT04541186/SAP_001.pdf